CLINICAL TRIAL: NCT04731831
Title: Characterization of Immunogenicity of Tumor Necrosis Factor Inhibitors in Arthritis Patients With Poorer Treatment Response Due to Gender, Obesity and Smoking Status.
Brief Title: Characterization of Immunogenicity of TNF Inhibitors in Arthritis Patients With Poorer Treatment Response.
Status: Recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Karen Buch Lauridsen, Principal Investigator, Aalborg University Hospital
Other Study IDs: N-20200063
Record Dates: First submitted 2020-12-19; First posted 2021-02-01 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA Whole Blood EDTA-plasma, EDTA-buffy coat, serum.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with arthritis starting infliximab or adalimumab: Patients with Rheumatoid Artritis, Psoriatic Arthritis, Anchylosing Spondylitis starting treament with infliximab or adalimumab

SUMMARY:
The aim of the study is to explore whether the influence of gender, tobacco smoking and obesity on treatment response in tumor necrosis factor inhibitors (TNFIs) can be explained by high degree of inflammation, human leucocyte antigen (HLA) type, autoantibodies, TNF and TNFI concentration and presence of ADA.

DETAILED DESCRIPTION:
Tumor necrosis factor inhibitors (TNFIs) have been uses with success since 1999 in Denmark in treatment of various inflammatory diseases, eg. rheumatoid arthritis (RA), Chrohn's disease, psoriasis, psoriatic arthritis (PsA) and ankylosing spondylitis (AS).

TNFIs block a central cytokine in the inflammatory process, tumor necrosis factor (TNF).

Because the drugs are large proteins, they are prone to trigger an immune response and elicit anti-drug antibodies(ADA).

Epidemiologic studies have revealed that groups of patients (women, tobacco smokers, obese patients) with inflammatory rheumatic diseases have a lower response to TNFIs. The reasons for this are not fully elucidated. The hypothesis is that immunogenicity and changed pharmacokinetic of TNFI are causes of the inferior response.

The investigators will carry out a prospective clinical studies of 120 arthritis patients (RA, PsA and AS) initiating treatment with adalimumab or infliximab. The patients will be followed for 12 months and will be registered in DANBIO as normal praxis. Blood samples will be collected at baseline, 2, 4 and 12 months or at termination of the treatment.

Genotypes, autoantibodies, inflammation markers, TNFI and ADA will be measured.

The aim of the study is to explore:

A: If differences between men and women with respect to different markers of inflammation, human leucocyte antigen (HLA), autoantibodies, TNFI concentration and presence of ADAs can explain the lower response and adherence to the treatment among women.

B: If differences between smokers and non-smokers with respect to different markers of inflammation, HLA, autoantibodies, TNFI concentration and presence of ADAs can explain the lower response and adherence to the treatment among patients with arthritis who smoke tobacco.

C: If differences between obese and normal weight patients with respect to different markers of inflammation, HLA, autoantibodies, TNFI concentration and presence of ADAs can explain the lower response and adherence to the treatment.

The study will contribute with new knowledge, which hopefully can make the treatment more personalized and efficient.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Diagnosed with RA, PsA or AS.
* Starting treatment with infliximab or adalimumab.
* Co- treatment with csDMARD or glucocorticoid is acceptable.
* No new bDMARD is initiated at the time of sampling.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at department of Rheumatology in Aalborg Universityhospital, Denmark. Other sites in Jutland, Denmark may be inkluded later.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment response | 12 months
  Changes in disease activity score according to the diagnose. A reduction in the disease activity score indicates a good treatment response.
  * Disease Activity Score 28 joints with C-reactive protein (DAS28-CRP)
  * Disease Activity in Psoriasis Arthritis (DAPSA)
  * Ankylosing Spondylitis Activity Score (ASDAS)
  * Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
  * Bath Ankylosin Spondylitis Functional Index (BASFI)

SECONDARY OUTCOMES:
Immunogenesity | 12 months
  Antibodies directed against infliximab or adalimumab. Concentration of anti-drug-antibodies
Drug koncentration | 12 months
  Plasma koncentration of infliximab or adalimumab
Concentration of markers of inflammation | 12 months
  C-reactive protein (CRP), IL1, .
Concentration of autoantibodies | Day 1
  ANA, ACPA, IgM-RF
HLA-type | Day 1
  Genomic determination of Human Leucocyte antigens

CONTACTS AND LOCATIONS:
Overall Officials: Lene Dreyer, MD, Prof., Principal Investigator — Department of Clinical Medicine, Aalborg University and Aalborg University Hospital
Locations (1):
- Department of rheumatology, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tracey D, Klareskog L, Sasso EH, Salfeld JG, Tak PP. Tumor necrosis factor antagonist mechanisms of action: a comprehensive review. Pharmacol Ther. 2008 Feb;117(2):244-79. doi: 10.1016/j.pharmthera.2007.10.001. Epub 2007 Oct 26. PMID 18155297
- [Background] Elliott MJ, Maini RN, Feldmann M, Kalden JR, Antoni C, Smolen JS, Leeb B, Breedveld FC, Macfarlane JD, Bijl H, et al. Randomised double-blind comparison of chimeric monoclonal antibody to tumour necrosis factor alpha (cA2) versus placebo in rheumatoid arthritis. Lancet. 1994 Oct 22;344(8930):1105-10. doi: 10.1016/s0140-6736(94)90628-9. PMID 7934491
- [Background] Steenholdt C, Bendtzen K, Brynskov J, Ainsworth MA. Optimizing Treatment with TNF Inhibitors in Inflammatory Bowel Disease by Monitoring Drug Levels and Antidrug Antibodies. Inflamm Bowel Dis. 2016 Aug;22(8):1999-2015. doi: 10.1097/MIB.0000000000000772. PMID 27135483
- [Background] van Schie KA, Hart MH, de Groot ER, Kruithof S, Aarden LA, Wolbink GJ, Rispens T. The antibody response against human and chimeric anti-TNF therapeutic antibodies primarily targets the TNF binding region. Ann Rheum Dis. 2015 Jan;74(1):311-4. doi: 10.1136/annrheumdis-2014-206237. Epub 2014 Oct 23. PMID 25342759
- [Background] Kalden JR, Schulze-Koops H. Immunogenicity and loss of response to TNF inhibitors: implications for rheumatoid arthritis treatment. Nat Rev Rheumatol. 2017 Nov 21;13(12):707-718. doi: 10.1038/nrrheum.2017.187. PMID 29158574
- [Background] Meroni PL, Valentini G, Ayala F, Cattaneo A, Valesini G. New strategies to address the pharmacodynamics and pharmacokinetics of tumor necrosis factor (TNF) inhibitors: A systematic analysis. Autoimmun Rev. 2015 Sep;14(9):812-29. doi: 10.1016/j.autrev.2015.05.001. Epub 2015 May 15. PMID 25985765
- [Background] Mould DR. The Pharmacokinetics of Biologics: A Primer. Dig Dis. 2015;33 Suppl 1:61-69. doi: 10.1159/000437077. Epub 2015 Sep 14. PMID 26367860
- [Background] Zandman-Goddard G, Peeva E, Shoenfeld Y. Gender and autoimmunity. Autoimmun Rev. 2007 Jun;6(6):366-72. doi: 10.1016/j.autrev.2006.10.001. Epub 2006 Nov 13. PMID 17537382
- [Background] Hojgaard P, Ballegaard C, Cordtz R, Zobbe K, Clausen M, Glintborg B, Kristensen LE, Dreyer L. Gender differences in biologic treatment outcomes-a study of 1750 patients with psoriatic arthritis using Danish Health Care Registers. Rheumatology (Oxford). 2018 Sep 1;57(9):1651-1660. doi: 10.1093/rheumatology/key140. PMID 29893926
- [Background] Chimenti MS, Triggianese P, Conigliaro P, Tonelli M, Gigliucci G, Novelli L, Teoli M, Perricone R. A 2-year observational study on treatment targets in psoriatic arthritis patients treated with TNF inhibitors. Clin Rheumatol. 2017 Oct;36(10):2253-2260. doi: 10.1007/s10067-017-3769-4. Epub 2017 Jul 31. PMID 28762060
- [Background] Kennedy NA, Heap GA, Green HD, Hamilton B, Bewshea C, Walker GJ, Thomas A, Nice R, Perry MH, Bouri S, Chanchlani N, Heerasing NM, Hendy P, Lin S, Gaya DR, Cummings JRF, Selinger CP, Lees CW, Hart AL, Parkes M, Sebastian S, Mansfield JC, Irving PM, Lindsay J, Russell RK, McDonald TJ, McGovern D, Goodhand JR, Ahmad T; UK Inflammatory Bowel Disease Pharmacogenetics Study Group. Predictors of anti-TNF treatment failure in anti-TNF-naive patients with active luminal Crohn's disease: a prospective, multicentre, cohort study. Lancet Gastroenterol Hepatol. 2019 May;4(5):341-353. doi: 10.1016/S2468-1253(19)30012-3. Epub 2019 Feb 27. PMID 30824404
- [Background] Gladman DD, Antoni C, Mease P, Clegg DO, Nash P. Psoriatic arthritis: epidemiology, clinical features, course, and outcome. Ann Rheum Dis. 2005 Mar;64 Suppl 2(Suppl 2):ii14-7. doi: 10.1136/ard.2004.032482. PMID 15708927
- [Background] Egeberg A, Kristensen LE, Thyssen JP, Gislason GH, Gottlieb AB, Coates LC, Jullien D, Gisondi P, Gladman DD, Skov L, Mallbris L. Incidence and prevalence of psoriatic arthritis in Denmark: a nationwide register linkage study. Ann Rheum Dis. 2017 Sep;76(9):1591-1597. doi: 10.1136/annrheumdis-2016-210963. Epub 2017 May 8. PMID 28483767
- [Background] Kvien TK, Uhlig T, Odegard S, Heiberg MS. Epidemiological aspects of rheumatoid arthritis: the sex ratio. Ann N Y Acad Sci. 2006 Jun;1069:212-22. doi: 10.1196/annals.1351.019. PMID 16855148
- [Background] Rifbjerg-Madsen S, Christensen AW, Christensen R, Hetland ML, Bliddal H, Kristensen LE, Danneskiold-Samsoe B, Amris K. Pain and pain mechanisms in patients with inflammatory arthritis: A Danish nationwide cross-sectional DANBIO registry survey. PLoS One. 2017 Jul 7;12(7):e0180014. doi: 10.1371/journal.pone.0180014. eCollection 2017. PMID 28686639
- [Background] Hojgaard P, Glintborg B, Kristensen LE, Gudbjornsson B, Love TJ, Dreyer L. The influence of obesity on response to tumour necrosis factor-alpha inhibitors in psoriatic arthritis: results from the DANBIO and ICEBIO registries. Rheumatology (Oxford). 2016 Dec;55(12):2191-2199. doi: 10.1093/rheumatology/kew326. Epub 2016 Sep 19. PMID 27651526
- [Background] Ternant D, Ducourau E, Perdriger A, Corondan A, Le Goff B, Devauchelle-Pensec V, Solau-Gervais E, Watier H, Goupille P, Paintaud G, Mulleman D. Relationship between inflammation and infliximab pharmacokinetics in rheumatoid arthritis. Br J Clin Pharmacol. 2014 Jul;78(1):118-28. doi: 10.1111/bcp.12313. PMID 24354889
- [Background] Ellulu MS, Patimah I, Khaza'ai H, Rahmat A, Abed Y. Obesity and inflammation: the linking mechanism and the complications. Arch Med Sci. 2017 Jun;13(4):851-863. doi: 10.5114/aoms.2016.58928. Epub 2016 Mar 31. PMID 28721154
- [Background] Perricone C, Versini M, Ben-Ami D, Gertel S, Watad A, Segel MJ, Ceccarelli F, Conti F, Cantarini L, Bogdanos DP, Antonelli A, Amital H, Valesini G, Shoenfeld Y. Smoke and autoimmunity: The fire behind the disease. Autoimmun Rev. 2016 Apr;15(4):354-74. doi: 10.1016/j.autrev.2016.01.001. Epub 2016 Jan 7. PMID 26772647
- [Background] Mattey DL, Brownfield A, Dawes PT. Relationship between pack-year history of smoking and response to tumor necrosis factor antagonists in patients with rheumatoid arthritis. J Rheumatol. 2009 Jun;36(6):1180-7. doi: 10.3899/jrheum.081096. Epub 2009 May 15. PMID 19447930
- [Background] Glintborg B, Hojgaard P, Lund Hetland M, Steen Krogh N, Kollerup G, Jensen J, Chrysidis S, Jensen Hansen IM, Holland-Fischer M, Hojland Hansen T, Nilsson C, Espesen J, Nordin H, Rasmussen Loft AG, Pelck R, Lorenzen T, Flejsborg Oeftiger S, Unger B, Jaeger F, Mosborg Petersen P, Rasmussen C, Dreyer L. Impact of tobacco smoking on response to tumour necrosis factor-alpha inhibitor treatment in patients with ankylosing spondylitis: results from the Danish nationwide DANBIO registry. Rheumatology (Oxford). 2016 Apr;55(4):659-68. doi: 10.1093/rheumatology/kev392. Epub 2015 Nov 30. PMID 26628579
- [Background] Hojgaard P, Glintborg B, Hetland ML, Hansen TH, Lage-Hansen PR, Petersen MH, Holland-Fischer M, Nilsson C, Loft AG, Andersen BN, Adelsten T, Jensen J, Omerovic E, Christensen R, Tarp U, Ostgard R, Dreyer L. Association between tobacco smoking and response to tumour necrosis factor alpha inhibitor treatment in psoriatic arthritis: results from the DANBIO registry. Ann Rheum Dis. 2015 Dec;74(12):2130-6. doi: 10.1136/annrheumdis-2014-205389. Epub 2014 Jul 25. PMID 25063827
- [Background] Kiely PD. Biologic efficacy optimization--a step towards personalized medicine. Rheumatology (Oxford). 2016 May;55(5):780-8. doi: 10.1093/rheumatology/kev356. Epub 2015 Sep 30. PMID 26424837
- [Background] Pouw MF, Krieckaert CL, Nurmohamed MT, van der Kleij D, Aarden L, Rispens T, Wolbink G. Key findings towards optimising adalimumab treatment: the concentration-effect curve. Ann Rheum Dis. 2015 Mar;74(3):513-8. doi: 10.1136/annrheumdis-2013-204172. Epub 2013 Dec 10. PMID 24326008
- [Background] Mulleman D, Meric JC, Paintaud G, Ducourau E, Magdelaine-Beuzelin C, Valat JP, Goupille P; Centre National de la Recherche Scientifique UMR 6239 GICC. Infliximab concentration monitoring improves the control of disease activity in rheumatoid arthritis. Arthritis Res Ther. 2009;11(6):R178. doi: 10.1186/ar2867. Epub 2009 Nov 25. PMID 19939280
- [Background] Ibfelt EH, Jensen DV, Hetland ML. The Danish nationwide clinical register for patients with rheumatoid arthritis: DANBIO. Clin Epidemiol. 2016 Oct 25;8:737-742. doi: 10.2147/CLEP.S99490. eCollection 2016. PMID 27822121
- [Background] Strand V, Balsa A, Al-Saleh J, Barile-Fabris L, Horiuchi T, Takeuchi T, Lula S, Hawes C, Kola B, Marshall L. Immunogenicity of Biologics in Chronic Inflammatory Diseases: A Systematic Review. BioDrugs. 2017 Aug;31(4):299-316. doi: 10.1007/s40259-017-0231-8. PMID 28612180
- [Background] Quistrebert J, Hassler S, Bachelet D, Mbogning C, Musters A, Tak PP, Wijbrandts CA, Herenius M, Bergstra SA, Akdemir G, Johannesson M, Combe B, Fautrel B, Chollet-Martin S, Gleizes A, Donnellan N, Deisenhammer F, Davidson J, Hincelin-Mery A, Donnes P, Fogdell-Hahn A, De Vries N, Huizinga T, Abugessaisa I, Saevarsdottir S, Hacein-Bey-Abina S, Pallardy M, Broet P, Mariette X; ABIRISK Consortium. Incidence and risk factors for adalimumab and infliximab anti-drug antibodies in rheumatoid arthritis: A European retrospective multicohort analysis. Semin Arthritis Rheum. 2019 Jun;48(6):967-975. doi: 10.1016/j.semarthrit.2018.10.006. Epub 2018 Oct 12. PMID 30420245
- [Background] Siljehult F, Arlestig L, Eriksson C, Rantapaa-Dahlqvist S. Concentrations of infliximab and anti-drug antibodies in relation to clinical response in patients with rheumatoid arthritis. Scand J Rheumatol. 2018 Sep;47(5):345-350. doi: 10.1080/03009742.2018.1433232. Epub 2018 Apr 27. PMID 29701536